CLINICAL TRIAL: NCT02648750
Title: A Stroke Self-Management Programme Delivered by Rehabilitation Assistants Within an Early Supported Discharge Service: A Feasibility Randomised Controlled Trial
Brief Title: Stroke Self-Management Delivered by Rehabilitation Assistants Within an Early Supported Discharge Service
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jenny Freeman (Other)
Responsible Party: Sponsor-Investigator, Jenny Freeman, Reader in Physiotherapy and Rehabilitation, University of Plymouth
Organization: University of Plymouth (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 177976
Record Dates: First submitted 2015-12-24; First posted 2016-01-07 (Estimated); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Stroke
Keywords: self-management; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehabilitation Assistant (Experimental): Bridges stroke self-management programme. Delivered by rehabilitation assistants. Participants will receive a minimum of 4 sessions over a 4-6 week period.
  Interventions: Behavioral: Bridges self-management programme
- Therapist (Active Comparator): Bridges stroke self-management programme. Delivered by registered stroke therapists (Occupational therapists or physiotherapists).
  Participants will receive a minimum of 4 sessions over a 4-6 week period.
  Interventions: Behavioral: Bridges self-management programme

INTERVENTIONS:
Behavioral: Bridges self-management programme — The Bridges self-management programme is based on self-efficacy principles. It includes a Bridges stroke workbook consisting of stroke survivors' experiences and strategies, with space to record and reflect on personal goals and achievements, which the practitioner will work through with the participant. The practitioner will also used strategies based on key principles of self-management during interactions with patients.

SUMMARY:
This feasibility study evaluates whether it is possible to run a larger scale study to investigate the use of a self-management programme with adults who have recently had a stroke. Half of the participants will receive support with self-management from stroke therapists, while the other half will receive it from rehabilitation assistants.

DETAILED DESCRIPTION:
Supporting self-management post-stroke is a key priority in healthcare policy, but not yet embedded into the provision of stroke rehabilitation. Barriers to implementation include time and resource. The feasibility of using the Bridges Stroke Self-Management Programme within an Early Supported Discharge Service and delivery by Rehabilitation Assistants is unknown.

The aim of this study was to evaluate key trial parameters to inform the protocol of a future definitive trial into the effectiveness of Bridges delivered by rehabilitation assistants within an Early Supported Discharge Service.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of new stroke
* Being referred to the ESD service
* Medically stable
* Able to give informed consent
* Can follow a two-stage command

Exclusion Criteria:

* Being discharged to a care home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline Stroke Self-Efficacy Scale at 6 weeks | Baseline and 6 weeks

SECONDARY OUTCOMES:
Change from baseline Modified Rivermead Mobility Index at 6 weeks | Baseline and 6 weeks
  Functional mobility
Change from baseline SIPSO at 6 weeks | Baseline and 6 weeks
  social integration
Change from baseline EQ5D at 6 weeks | Baseline and 6 weeks
  health-related quality of life
Change from baseline PHQ-9 at 6 weeks | Baseline and 6 weeks
  depression

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Freeman, PhD, Study Director — Plymouth University

IPD SHARING:
Plan to Share IPD: No